CLINICAL TRIAL: NCT01006369
Title: Autophagy and Anti-Angiogenesis in Metastatic Colorectal Carcinoma: A Phase II Trial of Hydroxychloroquine to Augment Effectiveness of XELOX-Bevacizumab. A Study of the Cancer Institute of New Jersey Oncology Group (CINJOG)
Brief Title: Hydroxychloroquine, Capecitabine, Oxaliplatin, and Bevacizumab in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elizabeth Poplin, MD, Professor of Medicine, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0220090022; CINJ-070806; P30CA072720 (NIH); 070806 (Other: Rutgers Cancer Institute of New Jersey)
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Results first posted 2021-03-11 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FOLFOX6 + Bevacizumab + Hydroxychloroquine (Experimental): Arm A: FOLFOX6 + Bevacizumab + Hydroxychloroquine: Bevacizumab will be administered intravenously 5 mg/kg in 100 cc Normal Saline every 14 days on day one.
  Drug: hydroxychloroquine hydroxychloroquine 200 mg po BID daily
  Interventions: Drug: hydroxychloroquine
- XELOX + Bevacizumab + Hydroxychloroquine (Experimental): Arm B: XELOX + Bevacizumab + Hydroxychloroquine: Bevacizumab will be administered intravenously 7.5 mg/kg in 100 cc Normal Saline every 21 days.
  Drug: hydroxychloroquine hydroxychloroquine 200 mg po BID daily
  Interventions: Drug: hydroxychloroquine

INTERVENTIONS:
Drug: hydroxychloroquine — hydroxychloroquine 200 mg po BID daily

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Hydroxychloroquine may help chemotherapy and bevacizumab work better and kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving hydroxychloroquine together with capecitabine, oxaliplatin, and bevacizumab works in treating patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the progression-free survival (PFS) of patients with metastatic colorectal carcinoma treated with hydroxychloroquine in combination with capecitabine, oxaliplatin, and bevacizumab and to compare this to a previously reported median PFS of 7.9 months.

Secondary

* To measure the overall response rate.
* To measure the duration of response for responding patients.
* To measure the disease-control rate (complete response, partial response, or stable disease for at least 2 courses).
* To document the safety and feasibility of this regimen in these patients.
* To develop surrogate biomarkers for autophagy detection in patient tissue specimens and to characterize the effects of hydroxychloroquine on autophagy in patients in vivo.

OUTLINE: This is a multicenter study.

Patients receive bevacizumab IV over 30-90 minutes and oxaliplatin IV over 2 hours on day 1. Patients also receive oral capecitabine twice daily on days 1-15 and oral hydroxychloroquine twice daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Peripheral blood and tumor tissue samples may be collected for biomarker and other laboratory studies.

After completion of study treatment, patients are followed up for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed colorectal carcinoma

  * Metastatic disease
* Measurable disease, defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension (longest diameter to be recorded) as > 20 mm by conventional techniques or > 10 mm by spiral CT scan
* Brain metastases allowed provided they have been treated and stable for > 4 weeks

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* AST/ALT ≤ 3 times upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 times ULN
* PT (INR) ≤ 1.5
* Creatinine < 1.5 times ULN
* Creatinine clearance ≥ 30 mL/min
* Urine protein:creatinine ratio < 1.0 OR < 1 g protein by 24-hour urine collection
* Not on dialysis
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception before, during, and for 4 weeks after completion of study treatment
* Prior non-colonic malignancies allowed provided there is no current clinical evidence of persistent or recurrent disease AND the patient is not on active therapy, including hormonal therapy
* No uncontrolled hypertension, defined as systolic BP > 150 mm Hg or diastolic BP > 90 mm Hg, despite antihypertensive medications
* No cardiac disease, including any of the following:

  * NYHA class III-IV congestive heart failure
  * Unstable angina (anginal symptoms at rest)
  * New onset angina (began within the past 3 months)
  * Myocardial infarction within the past 6 months
  * Uncontrolled arrhythmia
* No thrombolic or embolic events (e.g., cerebrovascular accident including transient ischemic attacks) within the past 6 months
* No serious non-healing wound, ulcer, or bone fracture
* No significant traumatic injury within the past 28 days
* No neuropathy ≥ grade 2
* No evidence of bleeding diathesis or coagulopathy
* No condition that would impair the patient's ability to swallow whole pills
* No malabsorption problem
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No known G-6PD deficiency
* No retinal or visual field changes from prior 4-aminoquinoline compound use
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to capecitabine or hydroxychloroquine
* No other concurrent serious systemic disorders (including active infections) that, in the investigator's opinion, would compromise the safety of the patient or compromise the patient's ability to complete the study

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy for metastatic disease, except for adjuvant therapy that was completed ≥ 6 months before the first evidence of metastasis
* More than 28 days since prior major surgical procedure or open biopsy
* No concurrent anticoagulation with warfarin

  * Concurrent low molecular weight heparin (or an equivalent drug) allowed
* No concurrent hydroxychloroquine for treatment or prophylaxis of malaria
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent St. John wort
* No other concurrent investigational or anticancer agents or therapies

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2015-08-06 (Actual); Study Completion 2016-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A. Moss, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (4):
- United States (4):
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New Jersey Medical School/The University Hospital Cancer Center, Newark, New Jersey

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through the Rutgers Cancer Institute of New Jersey of New Jersey Oncology Group. The study was open to accrual on 05/8/2009 and terminated on 04/27/2016.
Pre-assignment Details: We are reporting results on 38 eligible patients. Nine patients were not eligible for participation.
Groups:
- FOLFOX6 + Bevacizumab + Hydroxychloroquine: bevacizumab: Arm A: FOLFOX6 + Bevacizumab + Hydroxychloroquine: Bevacizumab will be administered intravenously 5 mg/kg in 100 cc Normal Saline every 14 days on day one
  Arm B: XELOX + Bevacizumab + Hydroxychloroquine: Bevacizumab will be administered intravenously 7.5 mg/kg in 100 cc Normal Saline every 21 days
  hydroxychloroquine: hydroxychloroquine 200 mg po BID daily
- XELOX + Bevacizumab + Hydroxychloroquine: bevacizumab: Arm A: FOLFOX6 + Bevacizumab + Hydroxychloroquine: Bevacizumab will be administered intravenously 5 mg/kg in 100 cc Normal Saline every 14 days on day one
  Arm B: XELOX + Bevacizumab + Hydroxychloroquine: Bevacizumab will be administered intravenously 7.5 mg/kg in 100 cc Normal Saline every 21 days
  XELOX regimen: Capecitabine will be started at a dose of 1,000 mg/m2/day bid po (total daily dose = 2,000 mg/m2) for 14 days (28 doses) of the 21 day cycle. This cycle will be repeated every 21 days. Oxaliplatin will be started at a dose of 130 mg/m2, in 250 ml of D5W over 2 hours given day 1 of each cycle. This cycle will be repeated every 21 days.
  hydroxychloroquine: hydroxychloroquine 200 mg po BID daily
Period: Overall Study
Arm/Group | FOLFOX6 + Bevacizumab + Hydroxychloroquine | XELOX + Bevacizumab + Hydroxychloroquine
Started | 13 | 25
Completed | 1 | 0
Not Completed | 12 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FOLFOX6 + Bevacizumab + Hydroxychloroquine | XELOX + Bevacizumab + Hydroxychloroquine | Total
Number analyzed (Participants) | 13 | 25 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 14 | 25
  >=65 years | 2 | 11 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 12 | 16
  Male | 9 | 13 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 11 | 24 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 11 | 18 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 25 | 38

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Computed Kaplan-Meier survival curve estimates for progression free survival (PFS) and compared to historical controls of median PFS of 240 days. Evaluated response using RECIST criteria every 12 weeks.
Time Frame: 6 years
Population: Subjects received FOLFOX6 or XELOX at physicians discretion with bevacizumab abd HCQ 200 mg po daily BID until progressive disease or intolerable side effects. Subjects were not analyzed by treatment assigned.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FOLFOX6 + Bevacizumab + Hydroxychloroquine
Number analyzed (Participants) | 38
days | 424 [214 to 619]

2. Secondary Outcome: Overall Response Rate
Description: Response rate was evaluated every 12 weeks using RECIST criteria. CR+PR+Stable= overall response
Time Frame: 6 years
Population: Subjects were assigned to FOLFOX6 or XELOX at physicians discretion and were analyzed as one group. Overall response rate was 75%
Measure: Number; unit: percentage of participants responding
Arm/Group | FOLFOX6 + Bevacizumab + Hydroxychloroquine
Number analyzed (Participants) | 38
percentage of participants responding | 75

3. Secondary Outcome: Overall Survival
Description: Computed using Kaplan-Meier survival curve estimates which were compared to historical controls (median overall survival) was 21.3 months (596).
Time Frame: 6 years
Population: Subjects were assigned to FOLFOX6 or XELOX at physician discretion and were analyzed together.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FOLFOX6 + Bevacizumab + Hydroxychloroquine
Number analyzed (Participants) | 38
days | 788 [652 to 788]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 128 days per patient.
Arm/Group | FOLFOX6 + Bevacizumab + Hydroxychloroquine | XELOX + Bevacizumab + Hydroxychloroquine
All-Cause Mortality (participants affected / at risk) | 11/13 | 14/25
Serious Adverse Events (participants affected / at risk) | 4/13 | 12/25
Other Adverse Events (participants affected / at risk) | 13/13 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFOX6 + Bevacizumab + Hydroxychloroquine (N=13) | XELOX + Bevacizumab + Hydroxychloroquine (N=25)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 2 (2) — Disease progression
Allergic reaction/hypersensitivity (General disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstruction, GI - colon (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal - other (specific) (Gastrointestinal disorders) | 0 (0) | 2 (2) — GI bleed
Dehydration (Gastrointestinal disorders) | 1 (1) | 1 (1)
Neuropathy: motor (Nervous system disorders) | 1 (1) | 2 (2)
Pain - chest wall (General disorders) | 0 (0) | 1 (1)
Potassium, serum low (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFOX6 + Bevacizumab + Hydroxychloroquine (N=13) | XELOX + Bevacizumab + Hydroxychloroquine (N=25)
Decreased hemoglobin (Blood and lymphatic system disorders) | 4 (4) | 9 (9)
Hemolysis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Immune hemolytic anemia, drug related hemolysis
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 4 (4) | 4 (4)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 13 (32) | 10 (10)
Platelets (Blood and lymphatic system disorders) | 4 (4) | 4 (4)
Hypertension (Cardiac disorders) | 3 (3) | 4 (4)
Insomnia (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 0 (0) | 16 (16)
Fever (General disorders) | 0 (0) | 4 (4) — In the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L
Weight loss (General disorders) | 2 (2) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 8 (8)
Anorexia (Gastrointestinal disorders) | 3 (3) | 4 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 17 (17)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) — Dysphagia (difficulty swallowing)
Nausea (Gastrointestinal disorders) | 3 (3) | 9 (9)
Dehydration (Gastrointestinal disorders) | 0 (0) | 4 (4)
Mucositis/stomatitis - oral cavity (Gastrointestinal disorders) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 7 (7)
Hemorrhage, pulmonary upper respiratory - nose (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Potassium, serum low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
ALT, SGPT (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
AST, SGOT (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Albumin, serum low (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Glucose, serum high (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Lipase (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Mood alteration - depression (Nervous system disorders) | 1 (1) | 0 (0)
Neurology - motor (Nervous system disorders) | 1 (1) | 1 (1)
Neuropathy - sensory (Nervous system disorders) | 4 (4) | 24 (24)
Pain (General disorders) | 6 (6) | 3 (3)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes